CLINICAL TRIAL: NCT04923087
Title: Impact of Auditory Stimulation in Eating Pleasure : Multicentric Study With Biscuits With Crunchy Texture vs Soft Texture in 100 Seniors Affected or at Risk of Presbyacusis
Brief Title: Impact of Auditory Stimulation in Eating Pleasure (EDERE 2021)
Acronym: EDERE 2021
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21odonto03
Record Dates: First submitted 2021-06-04; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Frailty; Malnutrition; Anorexia; Presbycusis; Edentulism Nos
MeSH Terms: conditions — Frailty; Malnutrition; Anorexia; Presbycusis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patient hospitalized in geriatrics or EHPAD: Subjects 65 years of age or older, hospitalized in geriatrics or EHPAD residents
  Interventions: Device: Compare the noise and pleasure of crunching between two hyperprotein nutritional supplements

INTERVENTIONS:
Device: Compare the noise and pleasure of crunching between two hyperprotein nutritional supplements — Validate the evaluation criteria "Do you hear the biscuit crunch?" and "Is it a pleasure?"

SUMMARY:
Background. Decreased taste and smell contribute to loss of appetite (anorexia), and the resulting protein-energy malnutrition increases the frailty of the elderly. The risk of falls, disability, infections and depression often requires them to be institutionalized. Elderly, undernourished and toothless patients often complain about the monotony of a soft, mixed-texture diet. In a previous study, some participants highlighted the pleasure of crunching cookies that have a solid texture that can be eaten in any dental condition. However, the age-related decrease in hearing (presbyacusis) is frequent and progressive from the age of 60. The hypothesis of this work is that older patients may perceive a crunchy food crunching in their mouth, despite presbycusis. If the hypothesis is verified, this would make geriatric caregivers aware of the possibility of diversifying the texture of food, in order to stimulate the pleasure of eating and increase the dietary intake in this population of patients who are often undernourished, dysphagic, edentulous and hearing impaired. The originality of this study is to share the expertise of geriatricians and specialists in mastication/swallowing (dental surgeon, speech-language pathologist), hearing (ENT doctor, hearing care professional) and nutrition (dietician).

Type of study. Type of study MR-004 "Research not involving the human person". Protocol. Compare the noise and pleasure of crunching between two hyperprotein nutritional supplements: a soft filled cookie (Nutra Cake™, Délical, France) and a crunchy cookie of the Breton type (Protibis™, Solidages, France). Blind study impossible: each subject will eat a cookie then the other in a random order and will be his own control. The tests will be performed without the possible hearing aids, but with or without the dentures according to the patient's preference. Indeed, some patients have dental prostheses that are no longer suitable for chewing, and that they wear only for aesthetics. Objective. Validate the evaluation criteria "Do you hear the biscuit crunch?" and "Is it a pleasure?" If so, encourage diversification with crunchy foods with a suitable texture, as well as dental and prosthetic rehabilitation of dependent elderly people.

ELIGIBILITY:
Inclusion Criteria:

Subjects 65 years of age or older, hospitalized in geriatrics or EHPAD residents.

Exclusion Criteria:

risk of false route when eating cookies, allergy to an ingredient in cookies

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects 65 years of age or older, hospitalized in geriatrics or living in a nursing home.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Perception of crunching despite presbycusis | a 10-min session
  Subjects will be invited to eat two types of protein-rich cookies : Protibis (Solidages, France) and Nautre Cake (Delical, France). "Do you hear the biscuit crunch?" question will be asked.

SECONDARY OUTCOMES:
Evaluation of plesure felt | a 10-min session
  After eating each type of cookies, "Is it a pleasure?" question will be asked

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France